CLINICAL TRIAL: NCT02001038
Title: Survey of Current Management of Orthopaedic Complications in Charcot Marie Tooth Disease Patients
Brief Title: Survey of Current Management of Orthopaedic Complications in CMT Patients
Status: Completed | Type: Observational
Sponsor: University College London Hospitals (Other)
Collaborators: National Hospital for Neurology and Neurosurgery, London (Unknown); University of Iowa (Other); Children's Hospital of Philadelphia (Other); University of Pennsylvania (Other); University of Rochester (Other); Dubowitz Neuromuscular Centre (Other); Sydney Children's Hospitals Network (Other); Carlo Besta Neurological Institute (Other); Johns Hopkins University (Other); Vanderbilt University (Other); University of Washington (Other); National Institutes of Health (NIH) (NIH); Stanford University (Other); Data Management and Coordinating Center (DMCC) (Other); Federal, State foundation and industry support: National Institute of Health (NIH), Muscular Dystrophy Association, Charcot Marie Tooth Association (Unknown)
Responsible Party: Principal Investigator, Prof Mary Reilly, Professor of Clinical Neurology and Consultant Neurologist, University College London Hospitals
Other Study IDs: INC 6608
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Charcot-Marie-Tooth Disease
MeSH Terms: conditions — Charcot-Marie-Tooth Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Orthopaedic surgeons: Orthopaedic surgeons who perform surgical procedures for foot deformities in CMT patients at participants centres.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey

SUMMARY:
Charcot-Marie-Tooth (CMT) disease is the most common inherited peripheral neuropathy. Foot deformities are frequent complications in CMT patients and orthopaedic surgery is often required. As yet there are no systematic studies on the management of orthopaedic complications in CMT patients and the current approach varies between centres. This study is a survey with the aim of understanding the current surgical approach to orthopaedic complications in CMT.

The target population includes orthopaedic surgeons who perform surgical procedures for foot deformities in CMT patients attending centres participating in the Inherited Neuropathies Consortium (INC).

DETAILED DESCRIPTION:
The study protocol consists of a survey addressed to orthopaedic surgeons. The survey will be completed once and it includes two different scenarios of typical CMT patients (one adult and one child).

The orthopaedic surgeons will be asked which surgical procedures they would apply to each scenario:

* forefoot cavus,
* clawtoes and
* hindfoot varus

No medications or therapeutic agents are a component of this project.

ELIGIBILITY:
Inclusion Criteria:

* Orthopaedic surgeons who perform surgical procedures for foot deformities in CMT patients attending centres participating in the Inherited Neuropatheis Consortium (INC)
* Willing to complete survey

Exclusion Criteria:

* Does not read or speak English
* Inability to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Orthopaedic surgeons who perform surgical procedures for foot deformities in CMT patients attending centres participating in INC.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2013-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Procedural correlations among orthopaedic surgeons on management of foot deformities in CMT patients | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Prof Mary Reilly, Study Chair — National Hospital for Neurology and Neurosurgery
Locations (1):
- National Hospital for Neurology and Neurosurgery, London, United Kingdom